CLINICAL TRIAL: NCT02994862
Title: One Year Clinical Evaluation of E. Max Laminate Veneers With and Without Using Galla Chinnesis as Natural Cross Linking and Remineralizing Agent Before Bonding to Teeth With Amelogenesis Imperfecta
Brief Title: E. Max Laminate Veneers With and Without Using Galla Chinnesis as Natural Cross Linking and Remineralizing Agent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Gamal Fahmy Mohammed, B.D.S, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1226500339
Record Dates: First submitted 2016-12-08; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Amelogenesis Imperfecta
MeSH Terms: conditions — Amelogenesis Imperfecta

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galla Chinnesis (Experimental): new Remineralizing Agent before Bonding to teeth with amelogenesis imperfecta
  Interventions: Other: Galla Chinnesis
- Conventional Bonding (Active Comparator): Normal Bonding Method
  Interventions: Other: Conventional Bonding

INTERVENTIONS:
Other: Galla Chinnesis — new Remineralizing Agent before Bonding to teeth with amelogenesis imperfecta
  Arms: Galla Chinnesis
Other: Conventional Bonding — Normal Bonding Protocol
  Arms: Conventional Bonding

SUMMARY:
In teeth requiring laminate veneers with amelogenesis imperfecta Will application of galla chinensis before Bonding of laminate veneers with adhesive resin cement provide better survival rate than conventional Bonding method

DETAILED DESCRIPTION:
one year Clinical evaluation of laminate veneers with amelogenesis imperfecta Will application of galla chinensis before Bonding of laminate veneers with adhesive resin cement provide better survival rate than conventional Bonding method

ELIGIBILITY:
Inclusion Criteria:

All subjects are required to be:

* From 18-60 years old, and able to read and sign the informed consent document.
* Physically and psychologically able to tolerate conventional restorative procedures
* Have no active periodontal or pulpal diseases, have teeth with good restorations
* Patients with teeth problems indicated for laminate veneer (e.g. discoloration, fracture not involve more than 50% enamel loss, mild malposition, ….)
* Willing to return for follow-up examinations and evaluation

Exclusion Criteria:

* Patients in the growth stage with partially erupted teeth
* Patient with fractured teeth of more than 50% enamel loss
* Patients with poor oral hygiene and motivation
* Pregnant women
* Psychiatric problems or unrealistic expectations
* Lack of opposite occluding dentition in the area intended for restoration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
marginal adaptation assessed by clinical evaluation using dental mirror and probe | 1 year
  clinical evaluation of marginal adaptation

SECONDARY OUTCOMES:
Patient satisfaction assessed using a Questionnaire | 1 Year
  Questionnaire for patient satisfaction

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cheng L, ten Cate JM. Effect of Galla chinensis on the in vitro remineralization of advanced enamel lesions. Int J Oral Sci. 2010 Mar;2(1):15-20. doi: 10.4248/IJOS10019. PMID 20690414